CLINICAL TRIAL: NCT00934063
Title: A 24-month Prospective, Non-interventional, Observational Study on the Composite Clinical Endpoint (GET-Score) Reflecting Quality of Life, Body Composition and Cholesterol Metabolism in Patients Treated With Norditropin® (Somatropin)
Brief Title: An Observational Study Validating a Score That Quantifies the Therapeutic Response to Treatment With Norditropin®
Acronym: GET
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3709
Record Dates: First submitted 2009-07-02; First posted 2009-07-08 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: somatropin
- B
  Interventions: Other: No treatment given

INTERVENTIONS:
Drug: somatropin — For s.c. (under the skin) injection. Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Groups: A
Other: No treatment given — Control group not receiving treatment
  Groups: B

SUMMARY:
This observational study is conducted in Europe. The aim of this observational study is to investigate the changes in a score (GET-score) which includes quality of life, body composition and cholesterol metabolism in patients on growth hormone treatment. The GET score stands for: Growth hormone deficiency and Efficacy of Treatment, and is a quantitative measurement of the efficacy of the treatment with growth hormone in adults.

ELIGIBILITY:
Inclusion Criteria:

* Severe acquired growth hormone deficiency
* No treatment with somatropin in the last 24 months before study participation
* Written informed consent

Exclusion Criteria:

* Contraindications for the treatment with somatropin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acquired growth hormone deficiency who have been deemed appropriate to receive Norditropin® as treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Improvement of an integrated score which consists of Quality of Life (QoL), body composition, lipid metabolism, bone mineral density | at 0, 3, 6, 12, 18 and 24 months after treatment initiation

SECONDARY OUTCOMES:
Health related quality of life (SF-36; EQ-5D) | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Disease related absences from work | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Bone mineral density DXA Z-score lumbar | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Total cholesterol, HDL, LDL | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Body composition: fat mass, fat-free mass, impedance (BIA) | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Waist-circumference | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Blood pressure | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Adverse Drug Reactions and Severe Adverse Drug Reactions | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Triceps skinfold thickness | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
Upper arm circumference | at 0, 3, 6, 12, 18 and 24 months after treatment initiation
IGF-I (Insulin-like growth factor 1) | at 0, 3, 6, 12, 18 and 24 months after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mainz, Germany

REFERENCES:
- [Derived] Kann PH, Bergmann S, Bidlingmaier M, Dimopoulou C, Pedersen BT, Stalla GK, Weber MM, Meckes-Ferber S. Design of the Growth hormone deficiency and Efficacy of Treatment (GET) score and non-interventional proof of concept study. BMC Endocr Disord. 2018 Feb 13;18(1):10. doi: 10.1186/s12902-018-0237-3. PMID 29433573
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com